CLINICAL TRIAL: NCT03635801
Title: The MyoVista Angiography Angioplasty Percutaneous Coronary Intervention - The MAAP Trial
Brief Title: The MyoVista Angiography Angioplasty Percutaneous Coronary Intervention Trial
Acronym: MAAP
Status: Terminated | Type: Observational
Why Stopped: Due to PI's unavailability
Sponsor: Royal Cornwall Hospitals Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2018.RCHT.53
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease; Diastolic Dysfunction
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MyoVista 12 Lead (ECG) NSTEMI: Patients enrolling in this clinical investigation will undergo a standard 12-lead ECG using the MyoVista 12-lead hs ECG device. An ECG is a quick, safe and painless test. No electricity is put into the body while it's carried out.
  There may be some slight discomfort when the electrodes are removed from the skin - similar to removing a sticking plaster - and some people may develop a mild rash where the electrodes were attached.
  An ECG is performed under controlled conditions.
  Interventions: Device: MyoVista 12 lead Electrocardiogram (ECG)

INTERVENTIONS:
Device: MyoVista 12 lead Electrocardiogram (ECG) — MyoVista 12 Lead Electrocardiogram (ECG)

SUMMARY:
Purpose of this clinical investigation: clinical evaluation/accuracy of HeartSciences MyoVista High-Sensitivity (hsECG) 12 lead Electrocardiogram device, for patients presenting with cardiac related chest pain and/or Non ST-segment Elevation Myocardial Infarction (NSTEMI). To assess the early intervention of N-STEMI patients. Determine if clinical outcomes can be improved. Assessment will be made on the MYOVISTA's indices, numerical values, and sensitivity/specificity for early detection of cardiac dysfunction/disease,i.e. Coronary Artery Disease (CAD). Primary objective to ascertain efficacy of the MyoVista and evaluate its usefulness in expediting patients that require further investigation/procedure by way of angiography, thus improving the patient care pathway. Recruitment will take place at the Royal Cornwall Hospitals Trust, the Sponsor who will fund the research. A single centre study. Participants will undergo a 12 lead MyoVista ECG in addition to a standard 12 lead ECG. This is not an invasive procedure and carries no risk to the patient. There will be no change in the patient care pathway. The study will last c. 2 years, enrolment of patients ceasing once the statistically significant number to power the study has been met which is sufficient and ethical. Prerequisites for inclusion to the clinical investigation include:

* Signed informed consent prior to any procedure relating to the investigation
* Patient compliance with the clinical investigational plan
* Follow-up appointment(s) attendance
* Patient(s) presenting to hospital with a clinical diagnosis of Non ST-segment Elevation Myocardial Infarction
* Notable Electrocardiogram morphological changes, consistent with Myocardial Ischaemia (MI) i.e. T-wave inversion, Biphasic T-wave, ST-segment depression
* Symptom onset of <12 hrs
* Elevated High Sensitivity Troponin Score
* GRACE score of >140 It is hoped that > 75% of patients seen will show willingness and compliance throughout the duration of the clinical investigation. Clinical benefits, early diagnosis of heart disease, streamlined triage of patients, reduction in morbidity/mortality, reduction in costs to National Health Service (NHS) and improved patient centered care.

DETAILED DESCRIPTION:
The purpose of this clinical investigation is the clinical evaluation and accuracy of HeartSciences MyoVista High-Sensitivity (hsECG) 12 lead Electrocardiogram devices, for patients presenting with cardiac chest pain and/or Non ST-segment Elevation Myocardial Infarction (NSTEMI). To assess the early intervention of N-STEMI patients and determine if clinical outcomes can be improved. In addition, assessment will be made on the MYOVISTA's indices, numerical values, and sensitivity/specificity for early detection of cardiac dysfunction/disease, namely Coronary Artery Disease (CAD). The Primary objective to ascertain efficacy of the MyoVista and evaluate its usefulness in expediting patients that require further investigation/procedure by way of angiography, thus improving the patient care pathway. This clinical investigation will answer an important clinical question, i.e. can outcomes in 'high-risk' N-STEMI patients be improved with the intervention of MyoVista 12 lead Electrocardiogram in the detection of heart disease/diastolic dysfunction, compared to current standard practice?This clinical investigation anticipates that outcomes are improved in 'high-risk' patients when early detection and diagnosis is made using the MyoVista. The clinical investigation should therefore determine whether there is a need for a change in patient management, specifically those patients presenting as N-STEMI. This will allow for earliest intervention, with the results and data of this clinical investigation informing National/International guidelines, practice and healthcare service provision. The Primary endpoint will be the acute reperfusion/revascularization of target coronary vessels by way of Percutaneous Coronary Intervention (PCI) with specified follow-up at six (6) and twelve (12) months, with twelve (12) month being the specified termination of the clinical investigation plan.This clinical investigation is a prospective, single-centred Pilot study. The total investigation duration is expected to be approximately 2 - 3 years.

ELIGIBILITY:
Inclusion Criteria: Inclusion Criteria

Prerequisites for inclusion to the clinical investigation will include:

* Signed informed consent prior to any procedure relating to the investigation
* Patient compliance with the clinical investigational plan
* Follow-up appointment(s) attendance
* Patient(s) presenting to hospital with a clinical diagnosis of Non ST-segment Elevation Myocardial Infarction
* Notable Electrocardiogram morphological changes, consistent with Myocardial Ischaemia (MI) i.e. T-wave inversion, Biphasic T-wave, ST-segment depression
* Symptom onset of <12 hrs
* Elevated High Sensitivity Troponin Score
* GRACE score of >140

Exclusion Criteria: Exclusion Criteria

* Have a recent documented Myocardial Infarction within 40 days prior to enrolment and commencement of this investigation
* Have had a recent Trans-Ischemic Attack (TIA) or Cerebrovascular Accident (CVA) within 3 months prior to enrolment and commencement of this investigation
* Have undergone cardiac surgery or coronary revascularisation within 3 months prior to enrolment and commencement of this investigation
* Be less than 18 years of age
* Involvement of vulnerable subjects (e.g. those lacking capacity to provide informed consent)
* Be pregnant or planning to become pregnant at commencement of this investigation
* Participation in another clinical investigational study. Justification for which is two fold - firstly, a conflict of interest between two clinical trials, and patient compliance. Use of drugs that may be contraindicated and alter the patient care pathway compromising the trial
* Have not provided a patient information sheet or patient consent form
* Any contraindication(s) to PCI
* Cardiogenic shock
* Awaiting Coronary Artery Bypass Grafting (CABG)
* Haemodynamic instability
* Recurrent Ventricular Tachycardia
* Recurrent Ventricular Fibrillation
* Atrial/Ventricular Septal defects (ASD's/VSD's)
* Those patients presenting with suspected N-STEMI and who are subsequently enrolled yet are deemed to have non-cardiac related chest pain post cardiological review will be discharged from the study and will therefore meet exclusion criteria. Neither further action nor participation will be expected
* N.B. In the event a patient is unable to make the decision to participate in the clinical investigation, i.e. lacking capacity to provide informed consent, then exclusion criteria will thus apply to such patients. For the purpose of this clinical trial, it is deemed that there will be no clinical benefit to either the patient nor the clinical investigation should inclusion of this cohort of patients be included and will be contrary to their quality of life.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non ST segment Myocardial Infarction (NSTEMI)
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
The MAAP Trial | Two Years
  The primary outcome is one that the MyoVista is a good predictor of the need for an Angiogram in those patients presenting with cardiac related chest pain, more specifically, NSTEMI patients. The Primary objective is to ascertain the efficacy of the MyoVista and evaluate its usefulness in expediting those patients that require further investigation/procedure by way of angiography/angioplasty, thus improving the patient care pathway.

SECONDARY OUTCOMES:
The MAAP Trial | Two Years
  The Secondary objective: To assess left ventricular function and ejection fraction, quality of life of patients, post procedure at 24 hours to asses any immediate benefit and with specified follow-up at six (6) and twelve (12) months, with twelve (12) month being the specified termination of the clinical investigation plan.
  Echocardiography, High Sensitivity Cardiac Troponin, CKD (Chronic Kidney Disease) cardiac markers will feature as further diagnostic tools in addition to the MyoVista and Angiography supporting in this clinical investigation. Assessment on significant improvement in left ventricular systolic function, ejection fraction, exercise tolerance and quality of life will be made at Six (6) and Twelve (12) months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Hadjiantoni, BSc Hons, Principal Investigator — Royal Cornwall Hospitals Trust
Locations (1):
- Royal Cornwall Hospital, Truro, Cornwall, United Kingdom